CLINICAL TRIAL: NCT04650048
Title: Modulation of an Experimental Prolonged Pain Model Using High Definition Transcranial Direct Current Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: Danish National Research Foundation (Other)
Responsible Party: Principal Investigator, Sebastian Kold Sørensen, Ph.D. fellow, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: N-20180085.p2
Record Dates: First submitted 2020-09-23; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Pain, Muscle; Healthy
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants are pseudo-randomly allocated to either the intervention or the control group so as the two groups are equally weighted on gender.
  Using the build in double-blind software of the HD-tDCS device, the participant as well as investigator is blinded to the protocol that is administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Both groups will receive an injection with 5 μg (0.5 ml) Nerve Growth Factor (NGF) in the first dorsal interosseous muscle (FDI muscle) prior to the HD-tDCS intervention. This injection a pain model, that is intended to induce muscle soreness and hyperalgesia.
  Interventions: Device: Active HD-tDCS
- Sham tDCS (Placebo Comparator): Both groups will receive an injection with 5 μg (0.5 ml) Nerve Growth Factor (NGF) in the first dorsal interosseous muscle (FDI muscle) prior to the HD-tDCS intervention. This injection a pain model, that is intended to induce muscle soreness and hyperalgesia.
  Interventions: Device: Sham HD-tDCS

INTERVENTIONS:
Device: Active HD-tDCS — Using the Starstim 32, HD-tDCS equipment we provide 20 minutes of 2 mA anodal multimodal stimulation of dorsolateral prefrontal cortex (DLPFC) and primary motor cortex simultaneously using ring-cathode configurations around the two anodes.
  Arms: Active tDCS
Device: Sham HD-tDCS — Using the Starstim 32, HD-tDCS equipment we provide sham stimulation with 30 seconds of ramping up to 2 mA intensity, then turning off for 19 minutes and then ramping down from 2 mA intensity to 0 in the last 30 seconds.
  This sham-configuration is intended to mimic the sensory experience of active HD-tDCS.
  Arms: Sham tDCS

SUMMARY:
The purpose of this double-blinded, parallel group randomized controlled trial is to investigate the effects of high definition transcranial direct current stimulation (HD-tDCS) on an experimental prolonged pain model in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this double-blinded, parallel group randomized controlled trial is to investigate the effects of high definition transcranial direct current stimulation (HD-tDCS) on an experimental prolonged pain model in healthy subjects. Forty healthy participants are administered the compound Nerve Growth Factor (NGF) in the right first dorsal interosseous muscle (FDI), which produced prolonged muscle soreness and hyperalgesia.

The forty participants are randomly allocated to either the control group receiving a Sham-tDCS paradigm, or the intervention group receiving three consecutive days of multimodal HD-tDCS targeting primary motor cortex (M1) and dorsolateral prefrontal cortex (DLPFC) simultaneously.

The somatosensory profile is assessed at baseline, before administration of NGF as well as prior and post each HD-tDCS session using standardised quantitative sensory testing.

It is hypothesised that the active HD-tDCS will modulate the neurological changes induced by the experimental pain condition, which will alleviate the hyperalgesia and hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women.
* Able to speak, read and understand English or Danish.

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Current use of opioids, antipsychotics, benzodiazepines
* Previous or current neurological, musculoskeletal, rheumatic, malignant, inflammatory or mental illnesses
* Current or prior chronic pain conditions
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-04-29 (Estimated)

PRIMARY OUTCOMES:
Change in pressure pain threshold. | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the pain thresholds are assessed before and after each intervention on the subsequent two days.
  A hand-held pressure algometer (Somedic, Hörby, Sweden) with a 1-cm2 probe will be used to record the pressure pain threshold. The pressure is increased gradually at a rate of 20 kPa/s. The measurement is repeated three times on the first dorsal interosseous muscle.
Change in pressure pain tolerance. | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the pain thresholds are assessed before and after each intervention on the subsequent two days.
  A hand-held pressure algometer (Somedic, Hörby, Sweden) with a 1-cm2 probe will be used to record the pressure pain threshold at baseline. The pressure is increased gradually at a rate of 20 kPa/s. The measurement is repeated three times on the first dorsal interosseous muscle. The participant is asked to rate the pain on a numerical rating scale (NRS) from 0-10. 0 representing no pain at all, and 10 representing the worst pain imaginable.

SECONDARY OUTCOMES:
Change in tactile detection threshold | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the sensory thresholds are assessed before and after each intervention on the subsequent two days.
  Tactile threshold will be measured using an anaesthesiometer consisting of a set of Von Frey filaments. The filaments are made of nylon fibre of various diameters so as to provide a range of forces of up to 300 grams. The minimum force that the subject can detect will be identified. This will be assessed on flexor carpi radialis on the right hand arm.
Change in mechanical pain threshold | Six assessments over three days: Baseline is assessed before any intervention at day one, and then the sensory thresholds are assessed before and after each intervention on the subsequent two days.
  Mechanical pain threshold (MPT) will be measured using a set of weighted pinprick stimulators with a flat contact area of 0.25 mm diameter that exert forces between 8 and 512 mN. Threshold procedures will use a method of limits with up to five series of ascending and descending stimulus intensities. This will be assessed on flexor carpi radialis on the right hand arm.
Change in conditioned pain modulation (CPM) | Three assessments over three days: Baseline is assessed before the stimulation at day one, and then again after the stimulation on the two subsequent days.
  A computer-controlled cuff pressure algometer (Nocitech, Denmark) with an air-filled tourniquet cuff (VBM, Germany) will be used to record cuff pressure-induced pain thresholds over the muscle bulk on the calfs. The pressure is increased gradually at a rate of 1 kPa/s to assess pain tolerance on a 0-10 VAS scale, where 0 is no pain at all and 10 is the worst pain imaginable.
  During CPM testing, the pain tolerance is first assessed on one leg marking the baseline. The pressure pain tolerance is then assessed on the same leg again, while the contralateral calf is applied a simultaneous painful pressure stimulus. The outcome of the CPM testing is the difference in pressure pain tolerance measured in kPA between the first and the second assessment. The larger the positive difference is between the baseline and the second assessment, the stronger CPM effect the subject has.
Change in temporal summation of pain (TSP). | Three assessments over three days: Baseline is assessed before the stimulation at day one, and then again after the stimulation on the two subsequent days.
  TSP will be applied using cuff pressure algometry. A total of 10 repeated mechanical pressure stimuli will be delivered at 0.5 Hz (1-s stimuli duration and 1-s interval between stimuli) to the test area. During the 10 repeated stimuli, subjects will continuously rate the pain intensity on a 10-cm continuous VAS. TSP is assessed on the calf of the right leg.
Change in electroencephalography response (EEG). | Three assessments over three days: The EEG will be recorded as a part of the HD-tDCS intervention.
  EEG will be recorded for four minutes prior to the HD-tDCS, during the HD-tDCS and four minutes immediately after the HD-tDCS. In the four minutes before and after HD-tDCS, the subject will have their eyes open for two minutes and their eyes closed for two minutes.
  The EEG data will be analyzed with a focus on the resting state. In particular the Alpha frequency brain waves are of interest, but exploratory analysis will be conducted on the Beta, Theta and Gamma frequency bands as well.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Graven-Nielsen, Prof., Principal Investigator — Aalborg University
Locations (1):
- Center for Neuroplasticity and Pain, Aalborg, North Denmark, Denmark